CLINICAL TRIAL: NCT04071652
Title: MATTERS Study - Mistral Percutaneous Tricuspid Valve Repair FIM Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mitralix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-475
Record Dates: First submitted 2017-04-13; First posted 2019-08-28 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Tricuspid Valve Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mistral (Experimental): The Mistral is an investigational device intended for percutaneous trans-catheter repair in high risk for surgery individuals suffering from functional Tricuspid Regurgitation (TR).
  The device system is to be used only in accordance with the approved Investigational Plan on subjects who have signed an informed consent form. Device use is limited to the approved study investigators.
  Interventions: Device: Mistral implantation

INTERVENTIONS:
Device: Mistral implantation — Mistral implant is implanted in the Tricuspid valve

SUMMARY:
The Mistral is an investigational device intended for percutaneous trans-catheter repair in high risk for surgery individuals suffering from functional Tricuspid Regurgitation (TR).

The device system is to be used only in accordance with the approved Investigational Plan on subjects who have signed an informed consent form. Device use is limited to the approved study investigators.

DETAILED DESCRIPTION:
The study is designed to clinically demonstrate device acute safety and technical performance (Primary Endpoints) along with longer FU device safety and effectiveness evaluation (Secondary Endpoint).

The main objectives of the study are :

* Evaluate the Acute safety of the implanted Mistral device post procedure and at 30 day follow up period.
* Evaluate the long term Safety of the device.
* Demonstrate effectiveness of the Mistral device in reducing TR.

Primary endpoints:

* Safety: Acute safety. Rate of device related SAE including device related mortality, stroke, MI, cardiac tamponade, surgery for failed percutaneous repair and non-elective cardiovascular surgery to treat an adverse event. At discharge and 30 days.
* Performance: Mistral Implantation rate of technical success (defined as successful device implantation with grasped chords from at least two leaflets.).

Secondary endpoints:

* Safety: Safety at 3, 6 and 12 months. Rate of device related SAEs at 3, 6 and 12 months.
* Effectiveness: TR reduction post-procedure, at discharge and 30 days, 3 and 6 months. Improved NYHA class, 6MWTdistance and KCCQ (quality of life) at 30 days, 3 and 6 months.

Relevant only for patients 11-20:

* Safety: Safety at 3, 6, 12 and 24 months. Rate of device related SAEs at 3, 6, 12 and 24 months.
* Effectiveness: TR reduction post-procedure, at discharge and 30 days, 3, 6, 12 and 24 months. Improved NYHA class, 6MWT distance and KCCQ (quality of Life) at 30 days, 3, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given signed study Informed Consent for participation prior to procedure.
* Subject is ≥ 18 years of age or legal age in host country
* Subject is willing and able to comply with all required follow-up evaluations
* Genders eligible for the study: Both genders
* Subject has TR of grade 3+ or more
* Subject has left ventricular ejection fraction (LVEF) >20 %
* Subject is of functional class 2 or more (NYHA)
* The subject is high risk to undergo TV surgery as assessed and consented by a cardiac surgeon and an interventional cardiologist at the site (center heart team), and according to ESC/EACTS guidelines on the management of valvular heart disease.
* Patients with Jugular and/or Femoral veins enabling catheterization with 12Fr catheters
* Life expectancy ≥ 1 year

Exclusion Criteria:

* Tricuspid Stenosis >mild
* Tricuspid Subvalvular calcification or calcification of the chordae.
* Subject has a history of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within the past 3 months.
* Subject has a history of a myocardial infarction (MI) in the past 3 months
* Subject has had a percutaneous interventional or other invasive cardiac or peripheral procedure ≤ 7 days of the index procedure
* Subject has a history of, or has active endocarditis
* Subject has echocardiographic evidence of intra-cardiac mass, thrombus, vegetation or soft-mobile deposits
* Subject is in acute pulmonary edema.
* Subject has hemodynamic instability requiring inotropic or mechanical support.
* Subject has a known hypersensitivity or contraindication to anticoagulant or antiplatelet medication
* Subject has renal insufficiency as evidenced by a serum Creatinine > 3.0mg/dL.
* Subject has ongoing infection or sepsis
* Subject has blood dyscrasias (leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis, or coagulopathy)
* Subject has an active peptic ulcer or has had gastrointestinal (GI) bleeding within the past 3 months prior to the index procedure
* Subject requires emergency surgery for any reason
* Subject has a known allergy to Nitinol alloys, 316L\304 stainless steel.
* Pregnant or lactating women.
* Patients being dependent upon the sponsor or upon the investigator or upon the investigational site.
* Subject has a known contrast media allergy
* Presence of high degree atrio-ventricular block (2nd or 3rd degree A-V block), or the presence of tri-fascicular block
* According to investigator on site the patient is suffering from a severe end stage disease (e.g. malignancy, severe pulmonary disease, liver disease, renal failure) and has a life expectancy of less than 1 year.
* Contraindication for treatment with dual antiplatelet therapy for at least 3 months
* Contraindication for TEE including trans-gastric views.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Safety: Acute safety. Rate of device related SAE | Until hospital discharge - up to 5 days post procedure day
  including device related mortality, stroke, MI, cardiac tamponade, surgery for failed percutaneous repair and non-elective cardiovascular surgery to treat an adverse event
Safety: Acute safety. Rate of device related SAE | At 30 days post procedure
  including device related mortality, stroke, MI, cardiac tamponade, surgery for failed percutaneous repair and non-elective cardiovascular surgery to treat an adverse event
Performance: Mistral Implantation rate of technical success | Procedure
  defined as successful device implantation with grasped chords from at least two leaflets

SECONDARY OUTCOMES:
Safety: Rate of device related SAE | at 3 months post procedure
Safety: Rate of device related SAE | at 6 months post procedure
Safety: Rate of device related SAE | at 12 months post procedure
Safety: Rate of device related SAE | at 24 months post procedure
  Relevant only for patients 11-20
Effectiveness: TR Grade reduction | post procedure (1 hour after implant device has been implanted)
Effectiveness: TR Grade reduction | Until hospital discharge - up to 5 days post procedure day
Effectiveness: TR Grade reduction | at 30 days post procedure
Effectiveness: NYHA class (categorization of heart failure extent) | at 30 days post procedure
Effectiveness: 6MWT distance | at 30 days post procedure
Effectiveness: KCCQ (Kansas City Cardiomyopathy Questionnaire) | at 30 days post procedure
Effectiveness: TR Grade reduction | at 3 months post procedure
Effectiveness: NYHA class (categorization of heart failure extent) | at 3 months post procedure
Effectiveness: 6MWT distance | at 3 months post procedure
Effectiveness: KCCQ (Kansas City Cardiomyopathy Questionnaire) | at 3 months post procedure
Effectiveness: TR Grade reduction | at 6 months post procedure
Effectiveness: TR Grade reduction | at 12 months post procedure
  Relevant only for patients 11-20
Effectiveness: TR Grade reduction | at 24 months post procedure
  Relevant only for patients 11-20
Effectiveness: NYHA class (categorization of heart failure extent) | at 6 months post procedure
Effectiveness: NYHA class (categorization of heart failure extent) | at 12 months post procedure
  Relevant only for patients 11-20
Effectiveness: NYHA class (categorization of heart failure extent) | at 24 months post procedure
  Relevant only for patients 11-20
Effectiveness: 6MWT distance | at 6 months post procedure
Effectiveness: 6MWT distance | at 12 months post procedure
  Relevant only for patients 11-20
Effectiveness: 6MWT distance | at 24 months post procedure
  Relevant only for patients 11-20
Effectiveness: KCCQ (Kansas City Cardiomyopathy Questionnaire) | at 6 months post procedure
Effectiveness: KCCQ (Kansas City Cardiomyopathy Questionnaire) | at 12 months post procedure
  Relevant only for patients 11-20
Effectiveness: KCCQ (Kansas City Cardiomyopathy Questionnaire) | at 24 months post procedure
  Relevant only for patients 11-20

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Haddassah, Jerusalem, Kiryat Hadassah
  - The Chain Sheba Medical Center at Tel HaShomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv